CLINICAL TRIAL: NCT07050134
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Efficacy and Safety of DR10624 in Patients With Hypertriglyceridemia and Carotid Atherosclerotic Plaque
Brief Title: A Trial to Evaluate the Efficacy and Safety of DR10624 in Patients With Hypertriglyceridemia and Carotid Atherosclerotic Plaque
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Junbo Ge (Other)
Collaborators: Zhejiang Doer Biologics Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Junbo Ge, Professor, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DR10624-203-01
Record Dates: First submitted 2025-06-05; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Hypertriglyceridemia; Carotid Atherosclerotic Plaques
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Referral and Consultation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DR10624 Injection (referred to as DR10624) (Active Comparator): The experimental group uses a titration administration method: starting with 12.5 mg QW for 4 weeks, then titrating to 25 mg QW for another 4 weeks, and finally increasing to 50 mg QW, which is maintained for 16 weeks, for a total of 24 doses.
  Interventions: Drug: DR10624 Injection；
- DR10624 Injection Placebo (referred to as placebo) (Placebo Comparator)
  Interventions: Drug: DR10624 Injection Placebo (referred to as placebo)

INTERVENTIONS:
Drug: DR10624 Injection； — The experimental group(Trial Drug)
  * Name: DR10624 Injection (referred to as DR10624)
  * Specification: 60mg (1mL)/vial
  * Active Ingredient: DR10624
  * Route of Administration: Subcutaneous injection
  * Packaging: Vial
  * Expiry Date: See the drug label
  * Storage Conditions: 2~8℃, protected from light
  * Manufacturer: Zhixiang Bio (Suzhou) Co., Ltd.
  * Supplier: Zhejiang Daor Biotechnology Co., Ltd.
  Arms: DR10624 Injection (referred to as DR10624)
Drug: DR10624 Injection Placebo (referred to as placebo) — (The control group)Placebo: Name: DR10624 Injection Placebo (referred to as placebo) Specification: 0mg (1mL)/vial (no active ingredient) Main Component: Normal saline Route of Administration: Subcutaneous injection Packaging: Vial Expiry Date: See the drug label Storage Conditions: 2~8℃, protected from light Manufacturer: Zhixiang Bio (Suzhou) Co., Ltd. Supplier: Zhejiang Daor Biotechnology Co., Ltd.
  Arms: DR10624 Injection Placebo (referred to as placebo)

SUMMARY:
This is a researcher-initiated study to evaluate the effect of DR10624 injection on carotid atherosclerotic plaques in patients with hypertriglyceridemia and carotid atherosclerotic plaques. The study adopts a randomized, double-blind, placebo-controlled design. The treatment group has one dose group, with titration administration. The administration starts at 12.5 mg QW for 4 weeks, then titrates to 25 mg QW for 4 weeks, and finally to 50 mg QW for 16 weeks, totaling 24 administrations. The control group receives placebo treatment with the same volume and administration method as the treatment group.

The study is divided into a screening period (3 weeks), a treatment period (24 weeks), and a follow-up period (4 weeks).

Screening period (W-3 to W-1):

Before participating in the screening, the subjects must fully understand all the risks and possible benefits of the trial and sign a written informed consent form voluntarily. Subjects entering the screening period will also receive therapeutic lifestyle guidance. Two fasting serum triglyceride tests are required during the screening period, with one test completed within one week before the first administration and an interval of at least one week between the two tests. On the day before the treatment period (D-1), eligible subjects will be randomly assigned and receive a randomization number.

Treatment period (W0 to W24):

Subjects who pass the screening will enter the treatment period and receive the target dose through titration. They will receive DR10624 injection at 12.5 mg QW or placebo QW for 4 weeks (W0 to W3), then at 25 mg QW or placebo QW for 4 weeks (W4 to W7), and finally at 50 mg QW or placebo QW for 16 weeks (W8 to W23), totaling 24 administrations over 24 weeks. Subjects need to return to the research center weekly for drug administration during W0 to W23. After each administration, injection site observations are required (30 minutes (±10 minutes) and 1 hour (±10 minutes) after each administration to check for injection site reactions), and corresponding efficacy and safety evaluations are completed as per the visit schedule. The last administration is on D162, and the end of treatment is defined as one week after the last administration (W24, D169). All subjects will return to the research center on D169 for the last efficacy and safety evaluations during the treatment period.

Safety follow-up period (W25 to W28):

All subjects who complete the treatment will enter a 4-week safety follow-up period. The final visit is on D197, and all subjects will return to the research center on D197 for the final assessment of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to sign the informed consent form before the start of any trial - related activities, with an understanding of the trial's procedures and methods, and a commitment to strictly adhere to the clinical trial protocol to complete the study.
2. Age between 18 and 65 years (not including 65 years), both male and female participants are acceptable.
3. Body Mass Index (BMI) of at least 24 kg/m² at the time of screening.
4. Two fasting triglyceride tests, spaced at least one week apart during the screening period, both showing results of at least 1.7 mmol/L but less than 5.7 mmol/L.
5. Confirmed carotid artery plaque: defined as a local structural change protruding into the carotid artery lumen, which is at least 0.5 mm or 50% greater than the surrounding carotid artery intima - media thickness (IMT), or IMT > 1.5 mm.
6. Carotid artery stenosis meets the following criteria: in asymptomatic individuals, less than 60%; in symptomatic individuals, less than 50% (by the NASCET method, see Appendix 2).
7. Ability to accept and comply with the therapeutic lifestyle interventions required by the protocol, and to maintain a stable lifestyle during the study period.

Exclusion Criteria:

1. Participants with a confirmed diagnosis of familial chylomicronemia syndrome (FCS) (Fredrickson Type I), apo CII deficiency, or familial dysbetalipoproteinemia (Fredrickson Type III); or participants with a high suspicion of the above three diseases.
2. Participants with a confirmed diagnosis of homozygous familial hypercholesterolemia.
3. Participants with type 1 diabetes mellitus (T1DM) or other types of diabetes; or participants with type 2 diabetes mellitus who are currently receiving hypoglycemic agents.
4. Participants with uncontrolled hypertension at screening, defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg despite medication.
5. Participants with a history of malignancy within five years prior to screening (excluding basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and cervical carcinoma in situ); or malignancy that occurred more than five years ago but is currently active.
6. Participants with a history of thyroid cancer, multiple endocrine neoplasia type 2, or a relevant family history.
7. Participants with clinically significant gastrointestinal motility disorders (e.g., severe diabetic gastroparesis), who have undergone or plan to undergo gastric bypass or gastric banding surgery during the study period, or who are on long-term use of drugs that directly affect gastrointestinal motility.
8. Participants with a history of acute pancreatitis within the past year, a history of chronic pancreatitis, or a symptomatic history of gallbladder disease (e.g., common bile duct stones, multiple gallstones, etc.) (excluding those who have undergone cholecystectomy).
9. A history of acute myocardial infarction, cerebral hemorrhage, or cerebral infarction (excluding lacunar infarction) before screening; hospitalization due to congestive heart failure, unstable angina pectoris, or transient ischemic attack; previous percutaneous coronary intervention or coronary artery bypass grafting or other cardiac surgery; or congestive heart failure classified as New York Heart Association (NYHA) functional class II or IV; or a history of carotid artery intervention.
10. Major surgery within 3 months prior to screening.
11. Participants with imaging evidence of diffuse carotid artery plaques, or two or more plaques in a single carotid artery.
12. Severe trauma or infection within 4 weeks prior to screening that has not yet resolved.
13. A history of severe active or unstable major depressive disorder (MDD) or other severe mental disorders (such as schizophrenia, bipolar disorder, or other severe mood or anxiety disorders), or a history of suicide attempt.
14. Known allergy to the study drug or its excipients, or a history of severe atopic diseases (such as asthma, urticaria, eczema, etc.) or severe allergic constitution (allergy to two or more foods or two or more drugs), or potential allergy to the study drug or its components or similar drugs.
15. Use of the following target drugs or participation in relevant clinical trials with experimental drugs within 3 months prior to screening, including drugs targeting glucagon - like peptide - 1 receptor (GLP - 1R), glucagon receptor (GCGR), and fibroblast growth factor 21 receptor (FGF21R).
16. Participation in other clinical trials and receipt of investigational drugs within 3 months prior to screening or within five half - lives of the investigational drug (whichever is longer).
17. Use of dipeptidyl peptidase - 4 (DPP - 4) inhibitors or participation in relevant clinical trials of DPP - 4 inhibitors and receipt of experimental drugs within 4 weeks prior to screening.
18. Use of lipid - lowering drugs or PCSK9 inhibitors (small interfering RNA class) within 4 weeks prior to screening.
19. Any of the following laboratory test results:

(1) ALT>3.0×upper limit of normal (ULN) and/or AST>3.0×ULN and/or TBIL>1.5×ULN; (2) Creatinine>1.5×upper limit of normal; or eGFR<45 mL/min/1.73m². (3) Serum calcium≥35 ng/mL (pg/mL); (4) TSH<lower limit of normal, or>10 U/ml; (5) Serum amylase or lipase>2.0×ULN; (6) Hb<110 g/L (male) or<100 g/L (female); (7) Positive HIV - Ab test; (8) HbA1c≥9.0% during screening. 20. Participants with any clinically significant 12 - lead electrocardiogram (ECG) abnormalities at screening:

1. Second - degree Mobitz II or third - degree atrioventricular block;
2. Long QT syndrome or QTcF>450 ms (male), QTcF>470 ms (female);
3. Other serious arrhythmias, such as paroxysmal supraventricular tachycardia, paroxysmal ventricular tachycardia, etc.

21. A history of drug abuse or excessive alcohol consumption within 3 months prior to screening. [Excessive alcohol consumption is defined as an average weekly intake of more than 21 units for men and more than 14 units for women (1 unit=360 mL beer, or 150 mL wine, or 45 mL spirits with 40% alcohol).] 22. Pregnant or breastfeeding women, or men or women with reproductive potential who are unwilling to use contraception throughout the study and for a specified period after the study ends [30 days after the last dose for women or 90 days for men].

23. Blood donation or blood loss of≥400 mL or platelet donation within 3 months prior to screening.

24. Participants with other factors that the investigator considers unsuitable for study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-05-11 (Estimated); Study Completion 2026-07-05 (Estimated)

PRIMARY OUTCOMES:
Change in carotid intima-media thickness (IMT) from baseline at treatment week 24 (W24). | 24weeks

SECONDARY OUTCOMES:
Change in IMT from baseline at W12 | 12weeks
Change in carotid plaque length from baseline at W12 and W24 | 12weeks，24weeks
Percentage change in carotid plaque area (TPA) from baseline at W12 and W24 | 12weeks，24weeks
Change in maximum carotid plaque thickness from baseline at W12 and W24 | 12weeks,24weeks
Change in carotid plaque ultrasound echo intensity from baseline at W12 and W24 | 12weeks and 24weeks
Change in VAP - detected lipoprotein subfraction analysis from baseline at W24 | 24weeks
Change in plasma concentration lysophosphatidylcholine and lysophosphatidylcholine from baseline at W12 and W24 | 12weeks and 24weeks
Percentage change in four blood lipid parameters (triglycerides, total cholesterol, LDL - C, HDL - C) from baseline at W12 and W24 | 12weeks and 24weeks
Safety evaluation | 28weeks
  Vital signs (body temperature)
Safety evaluation | 28weeks
  Vital signs ：Heart rate（beats per minute）
safety evaluation | 28weeks
  Vital signs ：blood pressure（mmHg）
safety evaluation | 28weeks
  Vital signs :respiratory rate (breaths per minute)
Number of participants with Physical examination | 28weeks
  Physical examination: including general appearance, skin and mucous membranes, head and neck, thyroid gland, chest and abdomen, spine and limbs, nervous system, and lymphatic system.
safety evaluation | 28weeks
  ECG：PR interval（ms）
safety evaluation | 28weks
  ECG:heart rate(bpm)
safety evaluation | 28weeks
  ECG:QT interval(ms)
safety evaluation | 28weeks
  ECG: QTcF(ms)
Number of Participants With Abnormal Laboratory Values | 28weeks
  Laboratory tests ： blood routine test（WBC、RBC、PLT、HGB、HCT、NEUT、BASO、EOS、MONO、LYM）； blood biochemistry test （ALT、AST、TBIL、DBIL、ALB、TP、GGT、ALP、LDH、K⁺、Na⁺、Ca²⁺、Cl-、P、UA、Urea/BUN、Cr、GLU、CK）； urine routine（pH、PRO、GLU、RBC、WBC、KET）
safety evaluation checklist | 28weeks
  Injection site reaction（Subcutaneous injection - the injection site is on both sides of the abdominal wall, more than 5cm away from the umbilicus.）

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, professor, Principal Investigator — Zhongshan Hospital Affiliated with Fudan University
Locations (1):
- Zhongshan Hospital Affiliated with Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boren J, Chapman MJ, Krauss RM, Packard CJ, Bentzon JF, Binder CJ, Daemen MJ, Demer LL, Hegele RA, Nicholls SJ, Nordestgaard BG, Watts GF, Bruckert E, Fazio S, Ference BA, Graham I, Horton JD, Landmesser U, Laufs U, Masana L, Pasterkamp G, Raal FJ, Ray KK, Schunkert H, Taskinen MR, van de Sluis B, Wiklund O, Tokgozoglu L, Catapano AL, Ginsberg HN. Low-density lipoproteins cause atherosclerotic cardiovascular disease: pathophysiological, genetic, and therapeutic insights: a consensus statement from the European Atherosclerosis Society Consensus Panel. Eur Heart J. 2020 Jun 21;41(24):2313-2330. doi: 10.1093/eurheartj/ehz962. No abstract available. PMID 32052833
- [Background] Touboul PJ, Hennerici MG, Meairs S, Adams H, Amarenco P, Bornstein N, Csiba L, Desvarieux M, Ebrahim S, Hernandez Hernandez R, Jaff M, Kownator S, Naqvi T, Prati P, Rundek T, Sitzer M, Schminke U, Tardif JC, Taylor A, Vicaut E, Woo KS. Mannheim carotid intima-media thickness and plaque consensus (2004-2006-2011). An update on behalf of the advisory board of the 3rd, 4th and 5th watching the risk symposia, at the 13th, 15th and 20th European Stroke Conferences, Mannheim, Germany, 2004, Brussels, Belgium, 2006, and Hamburg, Germany, 2011. Cerebrovasc Dis. 2012;34(4):290-6. doi: 10.1159/000343145. Epub 2012 Nov 1. PMID 23128470
- [Background] Liu Z, Peng Y, Li S, Lin Y, Huang Y, Chen W, Bao C, Zhou Z, Lin Z, Chen L. Increased circulating FGF21 level predicts the burden of metabolic demands and risk of vascular diseases in adults with type 2 diabetes. BMC Endocr Disord. 2023 Dec 7;23(1):272. doi: 10.1186/s12902-023-01523-y. PMID 38057786
- [Background] Conceicao-Furber E, Coskun T, Sloop KW, Samms RJ. Is Glucagon Receptor Activation the Thermogenic Solution for Treating Obesity? Front Endocrinol (Lausanne). 2022 Apr 25;13:868037. doi: 10.3389/fendo.2022.868037. eCollection 2022. PMID 35547006
- [Background] Cardona V, Ansotegui IJ, Ebisawa M, El-Gamal Y, Fernandez Rivas M, Fineman S, Geller M, Gonzalez-Estrada A, Greenberger PA, Sanchez Borges M, Senna G, Sheikh A, Tanno LK, Thong BY, Turner PJ, Worm M. World allergy organization anaphylaxis guidance 2020. World Allergy Organ J. 2020 Oct 30;13(10):100472. doi: 10.1016/j.waojou.2020.100472. eCollection 2020 Oct. PMID 33204386
- [Background] Zhang ZY, Hu CF, Wang MX, Lin J, Li JM, Wang RZ. Research on mechanism of PCS in damaging vascular endothelial cells and promoting formation of atherosclerosis via TLR4/TREM-1. Eur Rev Med Pharmacol Sci. 2018 Nov;22(21):7533-7542. doi: 10.26355/eurrev_201811_16295. PMID 30468503
- [Background] Navarese EP, Kolodziejczak M, Kereiakes DJ, Tantry US, O'Connor C, Gurbel PA. Proprotein Convertase Subtilisin/Kexin Type 9 Monoclonal Antibodies for Acute Coronary Syndrome: A Narrative Review. Ann Intern Med. 2016 May 3;164(9):600-7. doi: 10.7326/M15-2994. Epub 2016 Mar 22. PMID 26999484